CLINICAL TRIAL: NCT02338752
Title: Safety Issue and Efficacy Study of Combining Mix Vaccine and Standard Therapy in the Treatment of Pancreatic Carcinoma Patient
Brief Title: Safety and Efficacy Study of Mix Vaccine in Pancreatic Carcinoma Patient
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pancreatic cancer MV
Record Dates: First submitted 2015-01-11; First posted 2015-01-14 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2015-01

CONDITIONS: Pancreatic Neoplasms
Keywords: mix vaccine, pancreatic neoplasms, immunotherapy
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (Active Comparator): Patients in this group will be receiving standard therapy according to National Comprehensive Cancer Network (NCCN) guide line
  Interventions: Other: Standard Treatment
- MV+control (Active Comparator): Patients in this group will be receiving both standard therapy according to NCCN guide line and simultaneous injection of mix vaccine (MV).
  Interventions: Biological: MV; Other: Standard Treatment

INTERVENTIONS:
Biological: MV — MV is an intravenous intralipid suspension with 5 various vaccines, including DPT (diphtheria, pertussis, and tetanus ), typhoid, Staphylococcus aureus, paratyphoid A and B. Accessories include microbial A, lecithin, Twain-80, span 20 and soy-bean oil for injection. Inject 0.5 ml of the mixture subcutaneously every week. Best reaction after injection was defined as showing regional red and swollen at the injection point and mild fever and to achieve this, dose increasing or reduction is acceptable.
  Arms: MV+control
Other: Standard Treatment — Patient will receive a comprehensive histological and imaging check up to evaluate the histological type, stage of the disease and performance status. Then the patient will receive standard treatment, in brief, surgical resection for early stage patients and systemic treatment including chemotherapy for advanced stage patients, according to NCCN guide line.

SUMMARY:
The purpose of this study is to evaluate the safeness and effectiveness of mix vaccine (MV). Enrolled patients will receive standard treatment according to National Comprehensive Cancer Network (NCCN) guide line with or without combining MV injection. The efficacy and side effect will be compared between the two groups.

DETAILED DESCRIPTION:
In the study, after evaluation of the general and physical status, eligible patients will be enrolled and randomly assigned into two arms at an 1:1 ratio. In the control arm patients will be receiving standard therapy according to National Comprehensive Cancer Network (NCCN) guide line (control group) and in experimental arm, patients will be receiving simultaneous standard therapy and injection of mix vaccine (MV). MV will be injected weekly till disease progression.

Blood sample will be obtained at baseline and every week before MV injection for the assessment of clinical hematology, biochemistry measurements and immunology index (including immunoglobin, interleukin and interferon). Patients will be evaluated for toxicity throughout the study. Side effect, progression free survival, immunology index and general status will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients diagnosed with pancreatic carcinoma based on histology
* 2.Evaluable lesions on imaging study
* 3.Without known immunodeficiency
* 4.Age >18 and <80 years ago

Exclusion Criteria:

* 1.Patients is unable or unwilling to sign informed consent
* 2.Any autoimmune disorder, which is currently being treated with prednisone or any other immune suppressive medication
* 3.Positive HIV and/or RPR (rapid plasma reagin)
* 4.Female patient who is pregnant or breast feeding
* 5.Patients, based on the opinion pf the investigator, should not be enrolled into this study
* 6.Prior anti-cancer vaccine or biological immunotherapy
* 7.Allergic to any known ingredient of the MV compound

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
efficacy as measured by modified Response Evaluation Criteria In Solid Tumors (RECIST) criteria version 1.1 | 2 years

SECONDARY OUTCOMES:
safety as measured by Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 criteria | 1 month
immunology index | 2 years
  including lymphocyte subtype number and function, cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Kecheng Xu, MD, Study Chair — Fuda Cancer Hospital
Locations (1):
- Biological treatment center in Fuda cancer hospital, Guangzhou, Guangdong, China

REFERENCES:
- See also: related information — http://www.fudahospital.com/